CLINICAL TRIAL: NCT03281330
Title: Effect of Motor Entrainment to Auditory Cues and Music During Walking on Quality of Movement and Perceived Fatigue in Persons With Multiple Sclerosis (PwMS)
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: University Ghent (Other); Revalidatie & MS Centrum Overpelt (Other); National MS Center Melsbroek (Other)
Responsible Party: Principal Investigator, Peter Feys, prof. dr., Hasselt University
Other Study IDs: B67021629797
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- persons with Multiple Sclerosis
  Interventions: Behavioral: auditory cues and music during walking
- Healthy controls
  Interventions: Behavioral: auditory cues and music during walking

INTERVENTIONS:
Behavioral: auditory cues and music during walking — the effect of different conditions of auditory cueing and music on walking quality and perceived fatigue in persons with multiple sclerosis compared to healthy controls

SUMMARY:
The study investigates the effect of different conditions of auditory cueing and music on walking quality and perceived fatigue in persons with multiple sclerosis compared to healthy controls. The study extends over a four session period, each session lasting maximally 1h30 minutes The experimental conditions include participants walking to music and metronome (at different tempi) for 3minutes and 15 seconds per condition, with a rest period of 3 minutes in between each condition. Non-invasive equipment will be used. participants are equipped with sensors (watch-like straps at the wrists, ankles and across the chest) and are given wireless headphones.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MS of >1 year,
* no relapse in the last 1 month,
* ability to walk for 12 minutes without interruption,
* an average usual walking speed between the range of 0.4 and 1.2 m/s.

Exclusion Criteria:

* cognitive impairment hindering the understanding and execution of the experimental procedures
* pregnancy
* hearing impairment
* amusia
* beat deafness

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: persons with Multiple Sclerosis and healthy volonteers
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Spatio-temporal parameters of gait | day 1
  Participants wear portable APDM sensors. These sensors are activated during the walking, and record the spatio-temporal parameters of gait.
Spatio-temporal parameters of gait | week 1
  Participants wear portable APDM sensors. These sensors are activated during the walking, and record the spatio-temporal parameters of gait.
Spatio-temporal parameters of gait | week 2
  Participants wear portable APDM sensors. These sensors are activated during the walking, and record the spatio-temporal parameters of gait.
Spatio-temporal parameters of gait | week 3
  Participants wear portable APDM sensors. These sensors are activated during the walking, and record the spatio-temporal parameters of gait.
Parameter's of sychronisation | day 1
  Participants have two light ipods attached on their ankles- these are a part of the D-jogger system. The system is activated during the walking, and logs the synchronization parameters
Parameter's of sychronisation | week 1
  Participants have two light ipods attached on their ankles- these are a part of the D-jogger system. The system is activated during the walking, and logs the synchronization parameters
Parameter's of sychronisation | week 2
  Participants have two light ipods attached on their ankles- these are a part of the D-jogger system. The system is activated during the walking, and logs the synchronization parameters
Parameter's of sychronisation | week 3
  Participants have two light ipods attached on their ankles- these are a part of the D-jogger system. The system is activated during the walking, and logs the synchronization parameters

SECONDARY OUTCOMES:
subjective physical /mental fatigue | day 1
  After each experimental condition, the participant is asked 'how tired do you feel in your body on a scale of 0 to 10, 0 being not tired at all and 10 being exhausted'
subjective physical /mental fatigue | week 1
  After each experimental condition, the participant is asked 'how tired do you feel in your body on a scale of 0 to 10, 0 being not tired at all and 10 being exhausted'
subjective physical /mental fatigue | week 2
  After each experimental condition, the participant is asked 'how tired do you feel in your body on a scale of 0 to 10, 0 being not tired at all and 10 being exhausted'
physical /mental fatigue | week 3
  After each experimental condition, the participant is asked 'how tired do you feel in your body on a scale of 0 to 10, 0 being not tired at all and 10 being exhausted'
motivation | day 1
  he participants is asked: 'how motivating was it to walk to the last particular stimuli (in the metronome condition)/Song (in the music condition) on a scale of 0-5. ) being not motivating at all and 5 being very motivating'.
motivation | week 1
  he participants is asked: 'how motivating was it to walk to the last particular stimuli (in the metronome condition)/Song (in the music condition) on a scale of 0-5. ) being not motivating at all and 5 being very motivating'.
motivation | week 2
  he participants is asked: 'how motivating was it to walk to the last particular stimuli (in the metronome condition)/Song (in the music condition) on a scale of 0-5. ) being not motivating at all and 5 being very motivating'.
motivation | week 3
  he participants is asked: 'how motivating was it to walk to the last particular stimuli (in the metronome condition)/Song (in the music condition) on a scale of 0-5. ) being not motivating at all and 5 being very motivating'.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - University of Ghent, Ghent
  - Nationaal Multiple Sclerose Center, Melsbroek
  - Revalidatie & MS Centrum Overpelt, Overpelt

IPD SHARING:
Plan to Share IPD: Undecided